CLINICAL TRIAL: NCT00258791
Title: Effects of Pretreatment With Ibuprofen in Post- ECT Headache
Brief Title: Effects of Pretreatment With Ibuprofen in Post-Electroconvulsive Therapy (ECT) Headache
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: first postponed then cancelled as national drug authority changed requirements
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LVS-2005
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Mental Disorders
Keywords: Psychiatric disorders; ECT; Headache; Ibuprofen
MeSH Terms: conditions — Mental Disorders; Headache | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ibuprofen

SUMMARY:
The purpose of the study is to determine whether ibuprofen reduces post-ECT headache or reduces its severity.

DETAILED DESCRIPTION:
The aim of the study is to compare the severity of headache between patients who are receiving ibuprofen prior to ECT treatment with patients receiving placebo prior to ECT treatment.

Patients will be randomly assigned to receive either 600 mg ibuprofen 90 min prior to treatment or placebo orally, blinded to patient, physician and treatment team.

Patients will be asked about their headache with a visual analogue scale (VAS) 2 hours prior to and within 2 hours after treatment, 2-month, 6- month and 1 year follow-up [5].

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving ECT

Exclusion Criteria:

* Pregnancy, contraindications to ibuprofen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olav Morten Linaker, MD PhD, Principal Investigator — Norwegian University of Science and Technology